CLINICAL TRIAL: NCT03345576
Title: Testosterone and Long Pulse Width Stimulation for Denervated Muscles After Spinal Cord Injury
Brief Title: Testosterone and Long Pulse Stimulation After SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2649-R
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury
Keywords: Electric Stimulation; Spinal Cord Injuries; Muscle Denervation; carbohydrate metabolism; Lipids metabolism; Basal Metabolic Rate; Muscle Proteins; Mitochondria, Muscle; RNA; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be masked to the type of electrical stimulation (LPWS vs. standard NMES)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Testosterone and LPWS (Experimental): Twelve patients will undergo 1 year of supervised training examining the effects of testosterone replacement therapy (TRT) and long pulse width stimulation (LPWS) in persons with denervated spinal cord injury.
  Interventions: Device: Testosterone and LPWS
- Testosterone and standard NMES (Sham Comparator): Twelve patients will undergo 1 year of supervised training examining the effects of testosterone replacement therapy (TRT) and standard surface neuromuscular electrical stimulation (NMES) in persons with denervated spinal cord injury.
  Interventions: Drug: Testosterone and standard NMES

INTERVENTIONS:
Device: Testosterone and LPWS — Twelve patients will undergo 1 year of supervised training examining the effects of testosterone replacement therapy (TRT) and long pulse width stimulation (LPWS) in persons with denervated spinal cord injury.
  Other Names: Testosterone and long pulse width stimulation
  Arms: Testosterone and LPWS
Drug: Testosterone and standard NMES — Twelve patients will undergo 1 year of supervised training examining the effects of testosterone replacement therapy (TRT) and standard surface neuromuscular electrical stimulation (NMES) in persons with denervated spinal cord injury.
  Other Names: Testosterone and neuromuscular electrical stimulation
  Arms: Testosterone and standard NMES

SUMMARY:
Denervation following spinal cord injury (SCI) limits beneficial application of neuromuscular electrical stimulation (NMES). SCI with denervation results in extensive muscle atrophy that is accompanied with several cardio-metabolic health risks. The current proposal provides a novel intervention by examining the effects of long pulse width stimulation (LPWS) and testosterone replacement therapy (TRT) on restoring muscle size and leg lean mass after denervation in persons with SCI. This intervention will be rewarding for Veterans and Civilians with SCI who do not benefit from exercising their lower extremity muscles because denervation has limited the response to standard surface NMES. The investigators will study the biochemical mechanisms that contribute to changes in muscle size following this novel training. Combing both pharmaceutical and physical-therapeutic interventions will optimize restoration of muscle size after SCI.

DETAILED DESCRIPTION:
The long-term goal is to develop a rehabilitation strategy to mitigate the deleterious changes in muscle size and lower leg lean mass in persons with denervation following spinal cord injury (SCI). Currently, there is no available rehabilitation intervention following lower motor neuron (LMN) denervation. More than 46,000 Veterans are affected with SCI and may experience profound skeletal muscle atrophy and loss of lean mass and about 20-25% experience LMN denervation. Skeletal muscle cross-sectional area is 6 times smaller following LMN denervation compared to the innervated muscles. Denervation atrophy may be accompanied by several SCI health-related consequences.

Twelve weeks of twice weekly of surface neuromuscular electrical stimulation (NMES) resistance training (RT) can elicit more than a 35% increase in skeletal muscle size, decreased ectopic adipose tissue accumulation, increased insulin sensitivity after SCI. Moreover, the applicant's CDA-2 preliminary findings showed that 16 weeks of NMES-RT and testosterone replacement therapy (TRT) increased leg lean mass by 1.5 kg with no changes in the TRT group only. This was accompanied by an increase in the basal metabolic rate (BMR) of 218 kcal/day in the NMES-RT+TRT with no changes in the TRT group. During the course of recruitment for the study, 20% of individuals with SCI were excluded and could not benefit from exercising their lower extremity muscles, presumably because of LMN denervation.

Long pulse width stimulation (LPWS; 120-150 ms) has the potential to stimulate denervated muscles and to restore muscle size in people with SCI. The previous paradigm has focused on daily activation of the denervated muscles without applying progressive loading similar to RT. Daily training is not a clinically feasible approach in persons with SCI. Moreover, previous trials did not focus on enhancing the neuromuscular homeostasis by promoting the increase in lean mass independent of LMN denervation. Testosterone replacement therapy (TRT) has been shown to increase lean mass and basal metabolic rate in hypogonadal men with SCI. The investigators will determine if TRT+LPWS would increase skeletal muscle size, leg lean mass and improve overall metabolic health in SCI persons with LMN denervation. The investigators hypothesize that the one year TRT+LPWS protocol will upregulate protein synthesis pathways, down-regulate protein degradation pathways and increase overall mitochondrial health. Three specific aims will address these hypotheses. Aim 1 will assess the effects of TRT+LPWS compared to TRT+ standard neuromuscular electrical stimulation (NMES; as a control group) on the size of thigh skeletal muscle, intramuscular fat (IMF) and leg lean mass. Aim 2 will determine the association between the changes in skeletal muscle size, leg lean mass and the metabolic profile as determined by measuring BMR, serum lipids and carbohydrate profile. Aim 3 will investigate the cellular mechanisms responsible for evoking skeletal muscle hypertrophy following TRT+LPWS. This study is novel because it provides a feasible rehabilitation intervention by combining two approaches; which are likely to improve the quality of life in SCI persons with LMN denervation. If proven successful, the intervention will be easily translated into clinical practice for persons with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic motor complete SCI and level of injury of T10 and below
* Only participants with lower motor neuron (LMN) denervation as determined by EMG testing
* Participants must also have an absence of reflexes, denervation of both knee extensor muscles
* Tolerance to LPWS paradigm
* Both knee extensors will also have to be unresponsive (i.e., no observed tetanic contraction or twitches) to standard electrical stimulation procedures (stimulation frequency: 30 Hz; pulse duration:450 s and amplitude of the current:200 mA)
* All participants will undergo International Standards for Neurological Classification of SCI (ISNCSCI) examination for neurological level and function and only those with American Spinal Injury Classification (AIS A and B; i.e. motor deficit below the level of injury)

Exclusion Criteria:

* Diagnosis of neurological injury other than SCI
* Pre-existing medical conditions will be excluded (cardiovascular disease, uncontrolled type II DM and those on insulin requirements) or other concurrent medical conditions judged to be contraindicated by the site physician.
* Hematocrit above 50% and severe urinary tract infection or symptoms
* Those with hyper-physiological testosterone level above 800 ng/dl
* Those who will fail to tolerate the LPWS paradigm
* Progressive condition that would be expected to result in changing neurological status
* Lower extremity fracture around the knee joint (distal femur or proximal tibia) within the last 2 years from enrollment in the study
* Knee BMD < 0.60 gm/cm2
* Total hip BMD T-scores < -3.5
* Untreatable severe spasticity judged to be contraindicated by the site Physician
* Untreated or uncontrolled hypertension (systolic blood pressure >140 mmHg; diastolic blood pressure >90 mmHg)
* Pressure ulcer of the trunk, pelvic area, or lower extremities of grade 3 or more
* Psychopathology documentation in the medical record or history that may conflict with study objectives

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men with SCI, women will not be included in the current study because administering testosterone replacement therapy (TRT) is neither appropriate nor safe.
Enrollment: 12 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Gorgey, PhD PT, Principal Investigator — Hunter Holmes McGuire VA Medical Center, Richmond, VA
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The target audiences for dissemination of the results from this study include the VHA and its practitioners, the national SCI/D Services Office, the general healthcare community, and the Veteran population. The investigators will share findings with the SCI community. The SCI/D Services and PVA publish a quarterly newsletter that is sent to SCI practitioners across the VA system. The investigators will inform the VA community of the impact of these findings. The investigators will report findings to the scientific community via the American Congress of Rehab Medicine, American College of Sports Medicine and American Spinal Cord Injury Association (ASIA). The investigators will publish reports in different scientific journals.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Throughout the study and at the completion of the study.

REFERENCES:
- [Background] Gorgey AS, Khalil RE, Alrubaye M, Gill R, Rivers J, Goetz LL, Cifu DX, Castillo T, Caruso D, Lavis TD, Lesnefsky EJ, Cardozo CC, Adler RA. Testosterone and long pulse width stimulation (TLPS) for denervated muscles after spinal cord injury: a study protocol of randomised clinical trial. BMJ Open. 2022 Oct 5;12(10):e064748. doi: 10.1136/bmjopen-2022-064748. PMID 36198461
- [Result] Alazzam AM, Goldsmith JA, Khalil RE, Khan MR, Gorgey AS. Denervation impacts muscle quality and knee bone mineral density after spinal cord injury. Spinal Cord. 2023 Apr;61(4):276-284. doi: 10.1038/s41393-023-00885-3. Epub 2023 Mar 10. PMID 36899099

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant underwent a detailed history and physical exam by a certified study medical provider to ensure eligibility. This was followed by electrodiagnosis to ensure denervation of the knee extensor muscle groups.
Period: Overall Study
Arm/Group | Testosterone and LPWS | Testosterone and Standard NMES
Started | 6 | 6
Completed | 3 | 4
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone and LPWS | Testosterone and Standard NMES | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: Two participants withdrew after signing consent and being randomized without performing any intervention or study procedures.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 6 | 6 | 12
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two participants withdrew prior to performing any study procedures.
  years | 43 (12) | 47 (8) | 45 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants withdrew after signing consent forms without conducting any study procedures.
  Participants
    Female | 0 | 0 | 0
    Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Muscle Size Change
Description: Magnetic resonance imaging (MRI): The skeletal muscle area will be measured at baseline 6 months and 12 months after training (post-intervention).
Time Frame: Baseline, 6 months and 12 months
Population: We are reporting the results of magnetic resonance imaging analysis of the right whole thigh muscle cross-sectional area (CSA, cm^2) and knee extensor CSA (CSA, cm^2) at baseline, 6 months and 12 months of completion of Testosterone and LPWS or Testosterone and standard NMES.
Measure: Mean (Standard Deviation); unit: Muscle CSA (cm^2)
Arm/Group | Testosterone and LPWS | Testosterone and Standard NMES
Number analyzed (Participants) | 6 | 6
Muscle CSA (cm^2)
  Thigh Muscle CSA-BL (cm^2): number analyzed (Participants) | 4 | 5
  Thigh Muscle CSA-BL (cm^2) | 47.76 (12.76) | 31.1 (12.65)
  Whole Thigh Muscle CSA (cm^2) 6 months: number analyzed (Participants) | 4 | 5
  Whole Thigh Muscle CSA (cm^2) 6 months | 52.4 (16.7) | 36.0 (9.96)
  Whole Thigh Muscle CSA (cm^2) 12 months: number analyzed (Participants) | 2 | 4
  Whole Thigh Muscle CSA (cm^2) 12 months | 42.87 (22.4) | 41.1 (12.6)

2. Secondary Outcome: Basal Metabolic Rate
Description: Using indirect canopy after overnight 10-12 hours fast.
Time Frame: Baseline, 6 months and 12 months
Population: The numbers in P2 or at 12 months were different because of earlier withdrawal of participants from the study.
Measure: Mean (Standard Deviation); unit: Basal Metabolic Rate (BMR; Kcal/day)
Arm/Group | Testosterone and LPWS | Testosterone and Standard NMES
Number analyzed (Participants) | 5 | 5
Basal Metabolic Rate (BMR; Kcal/day)
  BMR-BL | 1634 (416) | 1580 (383)
  BMR- 6 Months | 1564 (428) | 1424 (250)
  BMR- 12 Months: number analyzed (Participants) | 2 | 3
  BMR- 12 Months | 1385 (182) | 1671 (194)

3. Secondary Outcome: Mitochondrial Complex Activities
Description: Performing a simple muscle biopsy and them muscle samples will be assayed to measure mitochondrial citrate synthase and other complexes.
Time Frame: Mitochondrial measurements were conducted over 1 year period at baseline [BL, before starting any intervention], Post-intervention 1 [ P1; 6 months after starting interventions] and Post-intervention 2 [P2-12 months after starting interventions]
Population: Three participants withdrew from Testosterone and LPWS before P2 as well as two participants withdrew from testosterone and standard NMES group before conducting P2.
Measure: Mean (Standard Deviation); unit: nmol/min/mg
Arm/Group | Testosterone and LPWS | Testosterone and Standard NMES
Number analyzed (Participants) | 5 | 5
nmol/min/mg
  Complex II-Baseline | 43 (63) | 46 (45)
  Complex II-Post-intervention 1 | 47 (39) | 36 (31)
  Complex II-Post-intervention 2: number analyzed (Participants) | 2 | 3
  Complex II-Post-intervention 2 | 14 (0.9) | 13 (10)

ADVERSE EVENTS:
Time Frame: through study completion during the entire course of the intervention until the end of the study or until withdrawal from the trial up to 12 months.
Arm/Group | Testosterone and LPWS | Testosterone and Standard NMES
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone and LPWS (N=6) | Testosterone and Standard NMES (N=6)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone and LPWS (N=6) | Testosterone and Standard NMES (N=6)
Skin irritations as result of using testosterone patches (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant reported skin irritation as result of using testosterone patches. Study medical provider recommended over the counter corticosteroid cream to reduce or decrease skin irritation. However, participant decided to withdraw from the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT03345576/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03345576/ICF_001.pdf